CLINICAL TRIAL: NCT05113472
Title: Adverse Reactions Following COVID-19 Vaccination: an Ecuadorian Experience
Brief Title: Adverse Reactions Following COVID-19 Vaccination Among Ecuadorian Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Respiralab (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-MED-001
Record Dates: First submitted 2021-11-08; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Adverse Drug Event
Keywords: adverse reactions; COVID-19; healthcare workers; Latin America; vaccination
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ecuadorian Healthcare Workers: All individuals involved were part of the first phase of the national COVID-19 vaccination plan in our country and were contacted through a local registry established by a local private university.
  Interventions: Biological: Pfizer-BioNTech COVID-19 vaccine

INTERVENTIONS:
Biological: Pfizer-BioNTech COVID-19 vaccine — Patients who were administered any dose of the Pfizer-BioNTech COVID-19 vaccine.

SUMMARY:
Limited large-scale studies have been conducted to investigate the adverse effects of COVID-19 vaccine in Latin America, particularly among the healthcare worker (HCW) population in Ecuador. The objective of this study was to assess a cohort of Ecuadorian healthcare workers for adverse reactions following vaccination with the Pfizer-BioNTech vaccine.

DETAILED DESCRIPTION:
The COVID-19 pandemic bears a burden on medical care and economies worldwide, however immunization at the population level provides a way for to reduce future morbidity and mortality. Vaccine hesitancy and reluctance in getting the COVID-19 vaccine and apprehensions about them have been present along the course of vaccination programs and mass immunizations across the world. Factors such as the quick, large-scale production of vaccines, lack of information, and uncertainty about adverse reactions in the public's eye as well about myths spreading through media channels have given rise to suspicion and fear in the Latin American population. Limited large-scale studies have been conducted to investigate the adverse effects of COVID-19 vaccine in Latin America, particularly among the healthcare worker (HCW) population in Ecuador. The objective of this study was to assess a cohort of Ecuadorian healthcare workers for adverse reactions following vaccination with the Pfizer-BioNTech vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Ecuadorian nationality
* Active practice in the medical field
* Received the Pfizer-BioNTech COVID-19 vaccine

Exclusion Criteria:

* Patients who voluntarily refused to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population included Ecuadorian healthcare workers who received the inoculation with the Pfizer-BioNTech COVID-19 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 1291 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Adverse reactions | 14 days since administration of either dose
  Pain, erythema, edema, pruritus, axillary edema, fever, cephalea, malaise, arthralgia, nausea, diarrhea, chills, fatigue, somnolence, syncope, paresthesia, anxiety, dizziness, epigastric pain, generalized rash, generalized pruritus, allergic rhinitis, petechiae, throat itchiness, allergic sinusitis, facial edema, bronchospasm, allergic conjunctivitis, dermatitis, eczema, ocular edema, urticaria, lip swelling, tongue swelling, facial rash, anaphylaxis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Espiritu Santo, Samborondón, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided